CLINICAL TRIAL: NCT07098780
Title: Role of Tranexamic Acid in Reducing Hemorrhagic Events in Bariatric Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Patel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Yusra Jamshed, Principal Investigator- Trainee General Surgery, Patel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH/IRB/2023/011
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhage; Bariatric Surgery; Obesity, Morbid
Keywords: Bariatric surgery; Tranexamic Acid; Hemorrhage in bariatric surgery; RCT; Randomised controlled trial
MeSH Terms: conditions — Hemorrhage; Obesity, Morbid | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transamine (Experimental): At the time of incision, 1000mg of the drug would be given intravenous, followed by two postoperative doses of 1000mg eight hours apart.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator)
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Tranexamic Acid — At the time of incision, 1000mg of the drug would be given intravenous, followed by two postoperative doses of 1000mg eight hours apart.
  Arms: Transamine
Other: Normal Saline (Placebo) — At the time of incision, 10ml of the drug would be given intravenous, followed by two postoperative doses of 10ml eight hours apart.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if tranexamic acid (TXA) helps reduce bleeding during bariatric surgery, such as laparoscopic sleeve gastrectomy (LSG) and mini gastric bypass (MGB). It will also look at how safe TXA is for people undergoing these procedures. The main questions it aims to answer are:

Does TXA reduce the amount of blood loss during bariatric surgery? Are there any side effects or complications in patients who receive TXA? Researchers will compare TXA to standard care (no TXA) to see if it is effective in reducing bleeding.

Participants will:

Receive either TXA or no TXA (placebo) before surgery Undergo standard bariatric surgery (LSG or MGB) Have their blood loss, hemoglobin levels, and any complications monitored during and after surgery

DETAILED DESCRIPTION:
STUDY BACKGROUND:

1. Introduction Obesity, over the past few decades, has become an area of concern as leading to major non-communicable diseases such as cardiovascular diseases, hypertension, type 2 diabetes mellitus, dyslipidemia and cancer. It has been declared a global epidemic by WHO due to the large prevalence of overweight and obese populations. A cross-sectional study conducted in Multan, Pakistan (2019) revealed the prevalence of obesity in women is 30.2% and in men at 24.3%. (1) Bariatric surgery remains an effective method of weight reduction in patients with obesity refractory to diet and drug therapy. Bariatric surgery has been established as a standard of treatment for morbid obesity. Laparoscopic Sleeve Gastrectomy (LSG) and Roux-en-Y Gastric bypass (RYGB) remain the two common surgical techniques. (2) These procedures are generally safe and effective, postoperative complications such as anastomotic leak, hemorrhage, obstruction, and Venous Thromboembolism (VTE) add to associated morbidities with up to 2% risk of serious complications, i.e., bleeding, leak etc. (3)

   Though the safety profile of LSG is superior to RYGB, bleeding still remains a significant morbidity peri-operative. (4) Available literature shows evidence of bleeding incidence to be 2-4%. (05) Hemorrhage in RYGB occurs roughly in 3% of the patients, (07) as compared to 2% in LSG. (08) These hemorrhagic events occur as staple line bleed, from mesenteric vessels and iatrogenic injury. () As hemorrhage leads to re-operation, various methods over time have been implied upon to reduce the risk of bleeding intra and post-operatively; these include suturing, buttressing, and human fibrin sealant.

   Where these techniques appear to be complicated and expensive, a cost-effective and simpler solution could be the use of Tranexamic acid (TXA). Tranexamic acid is a synthetic lysine analogue that blocks lysine binding sites on plasminogen molecules hence inhibiting the formation of plasmin, thereby inhibiting fibrinolysis. TXA is being successfully used for various gynecological, orthopedic, and cardiothoracic procedures. Its role in bariatric surgery is not very well established. (09) Data on the use of TXA in reducing peri-operative bleeding is not readily available. A prospective cohort on the effectiveness of reducing staple line bleeding in LSG patients suggests the use of TXA to be safe and cost-effective (10). Another retrospective study reported a reduction in staple line bleed by use of TXA (44 patients were given TXA post-operatively, and only 04 out of this required re-operation.) () A retro prospective cohort study conducted on 314 patients undergoing LSG infers that TXA administration at the time on induction reduces hemorrhagic incidents and rate of re-operations. (05) Data on randomized controlled trials investigating the role of TXA in patients undergoing LSG and MGB is not available.
2. OBJECTIVE:

   To determine the effectiveness of TXA in reducing hemorrhagic events when given prophylactically and post-operatively in patients undergoing LSG and MGB.
3. STUDY DESIGN:

This study is a multicenter (Patel hospital, Karachi and RIMS Trauma center) trial to evaluate the role of tranexamic acid in bariatric surgeries. The study is scheduled to be carried out, 6 months after the approval from ERC or till completions of sample size

1. INCLUSION CRITERIA:

   * Patients above 18 years of age AND
   * Undergoing Laparoscopic Sleeve Gastrectomy and MGB
   * Morbid obesity
2. EXCLUSION CRITERIA:

   * Patients on anti-platelets/anti-coagulants
   * Patients with inherited or acquired bleeding disorders
   * Patients with any acute medical condition predisposing to bleeding
   * Hormonal contraceptives
   * Known Allery to TXA
   * Female hormonal replacement therapy

   After screening subjects will be randomized.
3. RANDOMIZATION:

   Randomization will be carried out by block randomization technique. After randomization, the central research officer will instruct the pharmacy to dispense the drug/placebo in the standard dose. These doses will be given at the time of incision, and two more doses at intervals of eight hours
4. METHODOLOGY:

   Patients undergoing bariatric surgery would be evaluated on basis of inclusion/exclusion criteria and enrolled in study after written informed consent in Urdu/English At the time of incision, 1000mg of the drug would be given intravenous, followed by two postoperative doses of 1000mg eight hours apart.

   All of the procedures will be performed by the same surgeon. Patients undergoing the procedure will be given a prophylactic dose of S/C low molecular weight heparin for DVT prophylaxis 12 hours pre-operatively (40mg S/C for patients < 100kgs, 60mg S/C for patients >100kgs) and OD dose post-operatively for one week.

   Pre-operative hemoglobin will be checked/evaluated within 24 hours, while postoperative within 8 to 16 hours.

   Table 1: administration regime:

   TIME FRAME DOSE At the time of incision 1000mg IV route Post operative two doses 8 hours apart 1000mg IV route
5. PROCEDURE TECHNIQUE:

   LAPAROSCOPIC SLEEVE GASTRECTOMY:

   • -Pneumo peritoneum is created through Palmar's point, other ports are inserted under vision.

   • -Gastro esophageal junction is identified; greater curvature of stomach is mobilized till left crus of diaphragm superiorly and 3cms from pylorus inferiorly

   • -Stomach tube is created with stapler

   • -Leak test is performed

   • -Sheath and skin incisions are closed

   MINI-GASTRIC BY PASS

   • Pneumo peritoneum is created through Palmar's point, other ports are inserted under vision.

   • Dissection is done at crow's foot to enter lesser sac

   • Stomach tube is created with one transverse and four longitudinal staplers

   • Greater omentum is transected up to transverse colon
   * Antecolic, isoperistaltic side to side anastomosis is made using stapler, gastrotomy/enterotomy is closed using PDS 2/0 in continuous fashion
   * Leak test is performed
   * Skin is closed

     4. STUDY ASSESMENT:

<!-- -->

1. PRIMARY OUTCOMES:

   * Use of number of clips intraoperatively
   * Staple line over sewing
   * A drop in baseline hemoglobin
   * Need for intervention (endoscopy or re-operation)

     5. SAFETY ASSESMENT:

Patients who will require post operative TXA due to an uncontrolled hemorrhagic event, will be unblinded as intention to treat analysis

6. DATA MANAGEMNT:

In this study the study data will be collected by General Surgery resident in a Performa.

1) DETERMINATION OF SAMPLE SIZE:

Sample size is calculated by using the WHO sample size calculator and the following parameters were achieved.

Level of significance (α): 5 Power (1-β): 80 Test value of population proportion (P0): 0.108 Anticipated value of population proportion (Pa): 0.223 Sample size (n): 70 in each arm

2) SAMPLING TECHNIQUE:

Non-probability consecutive sampling is used.

2) STATISTICAL ANALYSIS

Data will be collected and analyzed by using SPSS version 22. Using descriptive statistics, qualitative data will be reported in percentages and frequencies.

Depending upon the distribution of data for continuous variables, the mean ± standard deviation or median ± interquartile range will be reported.

To check the distribution we will apply Shapiro Kolmogroove test on number of clips used, number of sutures used, Blood product transfusions, change in hemoglobin.

To check the significance level chi square test will be applied between categorical variables, Staple line over sewing, anastomotic leak (evident by melena or hematemesis), readmissions, and endoscopy, re operation with comparison TXA / Non TXA group.

For continuous variables Number of clips used, number of sutures used, Blood product transfusions, change in hemoglobin with TXA/ Non TXA group the student t-test or Mann Whitney U test will be applied.

Confounders will be adjusted by logistics regression or liner regression analysis.

Patients who will require post-operative TXA due to an uncontrolled hemorrhagic event, will be unblinded as intention to treat analysis.

A P-value <0.05 less

7. QUALITY DATA ASSURANCE: The investigator is responsible for verifying that data entries are accurate and correct by physically signing the Performa. Accurate documentation (source document) that supports the date entered in the Performa should be maintained.

The dosing date and time of investigational product/ placebo and any deviation from protocol procedures will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age AND
* Undergoing Laparoscopic Sleeve Gastrectomy and MGB
* Morbid obesity

Exclusion Criteria:

* Patients on anti-platelets/anti-coagulants
* Patients with inherited or acquired bleeding disorders
* Patients with any acute medical condition predisposing to bleeding
* Hormonal contraceptives
* Known Allery to TXA
* Female hormonal replacement therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Need for additional intervention intra operative after administration of transamine | From enrollment to 24 hours after surgical procedure
  Bleeding event intraoperative Use of clips intraoperatively Staple line over sewing A drop in baseline hemoglobin in 24 hours Need for intervention post operative 24 hours (endoscopy or re-operation)

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Murtaza, MBBS, FCPS, MRCS, MSc (epi), Study Director — Patel Hospital
Locations (1):
- Patel Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
These participants are patients of Patel Hospital, and none of their data will be shared anywhere outside hospital or the department. In department participants are known to on duty doctors, but no data is shared or will be shared to unauthorized personnel

REFERENCES:
- [Background] Klaassen RA, Selles CA, van den Berg JW, Poelman MM, van der Harst E. Tranexamic acid therapy for postoperative bleeding after bariatric surgery. BMC Obes. 2018 Dec 3;5:36. doi: 10.1186/s40608-018-0213-5. eCollection 2018. PMID 30524741
- [Background] Chakravartty S, Sarma DR, Chang A, Patel AG. Staple Line Bleeding in Sleeve Gastrectomy-a Simple and Cost-Effective Solution. Obes Surg. 2016 Jul;26(7):1422-8. doi: 10.1007/s11695-015-1986-y. PMID 26694209
- [Background] Zafar SN, Miller K, Felton J, Wise ES, Kligman M. Postoperative bleeding after laparoscopic Roux en Y gastric bypass: predictors and consequences. Surg Endosc. 2019 Jan;33(1):272-280. doi: 10.1007/s00464-018-6365-z. Epub 2018 Sep 19. PMID 30232617
- [Background] Augustin T, Aminian A, Romero-Talamas H, Rogula T, Schauer PR, Brethauer SA. Reoperative Surgery for Management of Early Complications After Gastric Bypass. Obes Surg. 2016 Feb;26(2):345-9. doi: 10.1007/s11695-015-1767-7. PMID 26140855
- [Background] https://link.springer.com/article/10.1007/s00423-022-02630-5
- [Background] Wolfe BM, Kvach E, Eckel RH. Treatment of Obesity: Weight Loss and Bariatric Surgery. Circ Res. 2016 May 27;118(11):1844-55. doi: 10.1161/CIRCRESAHA.116.307591. PMID 27230645
- [Background] Asif M, Aslam M, Altaf S, Atif S, Majid A. Prevalence and Sociodemographic Factors of Overweight and Obesity among Pakistani Adults. J Obes Metab Syndr. 2020 Mar 30;29(1):58-66. doi: 10.7570/jomes19039. PMID 32045513